CLINICAL TRIAL: NCT07020338
Title: Effects of Yoga on Menstrual Symptoms, Pain, Sleep Quality, and Aerobic Endurance in Young Women With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Yoga Effects in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Seda Uluşahin, PT PhD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-510
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary dysmenorrhea; Yoga; Menstrual symptoms; Sleep quality; aerobic endurance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group randomized controlled trial design. Participants were randomly assigned to either a yoga intervention group or a control group in a 1:1 ratio. Each participant remained in their assigned group for the entire study duration, and there was no crossover between groups. The outcome assessor was blinded to group allocation (single-blind design).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Intervention (Experimental): Participants in this group received a structured yoga program consisting of 50-minute sessions, twice per week, over three menstrual cycles.
  Interventions: Other: Yoga Exercise Program
- Control Group (No Intervention): Participants in this group received no intervention during the study period but were offered the yoga program after completion of the study.

INTERVENTIONS:
Other: Yoga Exercise Program — Participants in the intervention group received a structured yoga-based exercise program consisting of 50-minute sessions, conducted twice per week over a period of approximately 10-12 weeks (three menstrual cycles). The program was based on Hatha Yoga principles
  Arms: Yoga Intervention

SUMMARY:
The goal of this clinical trial was to assess whether a yoga-based exercise program could improve aerobic endurance, sleep quality, and reduce menstrual symptoms and pain in young women aged 18-25 with primary dysmenorrhea.

The main questions it aimed to answer were:

Did yoga reduce menstrual pain and symptom severity?

Did yoga improve sleep quality and aerobic endurance?

Researchers compared a yoga intervention group to a control group to determine whether the yoga program led to improvements in these outcomes.

Participants:

Were randomly assigned to either a yoga group or a control group

Completed assessments of menstrual pain (VAS), menstrual symptoms (Menstrual Symptom Scale), sleep quality (Sleep Diary), and aerobic endurance (Incremental Shuttle Walk Test and Endurance Shuttle Walk Test)

In the intervention group, attended 50-minute yoga sessions twice a week for three menstrual cycles

Participants in the control group were offered the same yoga program after the study period.

DETAILED DESCRIPTION:
Primary dysmenorrhea, defined as painful menstruation without an identifiable pelvic pathology, is one of the most prevalent gynecological conditions among young women, affecting up to 90% of this population. It is typically characterized by cramping lower abdominal pain, often accompanied by back or thigh discomfort, and may be associated with systemic symptoms such as nausea, fatigue, and gastrointestinal disturbances. These symptoms can impair daily functioning, reduce sleep quality, and limit physical activity and endurance. While pharmacologic treatments remain first-line therapy, non-pharmacologic, low-risk, and accessible interventions such as yoga have gained attention for their potential holistic benefits.

This randomized controlled trial was designed to evaluate the effects of an 8-week structured yoga program on aerobic endurance, sleep quality, menstrual pain, and menstrual symptom severity in young women with primary dysmenorrhea.

A total of 32 female participants, aged 18-25 years, who had reported primary dysmenorrhea with menstrual pain intensity greater than 40 mm on the Visual Analog Scale (VAS) for at least the past 6 months, were recruited and randomly assigned to either a yoga intervention group (n = 16) or a control group (n = 16). Participants were recruited through convenience and snowball sampling methods via social media and community announcements. Exclusion criteria included regular physical exercise, irregular menstrual cycles, pregnancy, prior childbirth, pelvic surgery, or use of hormonal or psychiatric medications.

The yoga program was delivered twice weekly in 50-minute sessions for 8 weeks (across three menstrual cycles). It included:

Asanas (postures) targeting flexibility and pelvic mobility

Pranayama (breathing exercises) aimed at autonomic regulation

Relaxation and mindfulness components to reduce stress and improve sleep

All participants underwent assessments at three timepoints (baseline, after menstrual cycle 1, and after menstrual cycle 3), specifically during the first 3 days of their menstruation.

Outcome Measures:

Pain intensity: assessed via Visual Analog Scale (VAS)

Menstrual symptoms: evaluated using the Menstrual Symptom Questionnaire (MSQ)

Attitudes toward menstruation: measured through the Menstrual Attitude Questionnaire (MAQ)

Sleep quality: assessed with a Sleep Diary, capturing both quantitative sleep parameters and subjective quality

Aerobic endurance: measured using two field tests:

Incremental Shuttle Walk Test (ISWT) - to evaluate maximum aerobic capacity

Endurance Shuttle Walk Test (ESWT) - to assess submaximal endurance at 70-85% VO₂peak

Each test included pre- and post-assessment of vital signs (heart rate, oxygen saturation, blood pressure) and perceived exertion (Modified Borg Scale). Testing was stopped according to safety thresholds (e.g., failure to match the pace, HR >85% max, or participant-reported symptoms).

The primary hypothesis was that the yoga group would show statistically significant improvements in sleep quality and aerobic endurance, and reductions in menstrual pain and symptom severity, compared to the control group.

This study aimed to contribute to the growing body of evidence supporting yoga as a safe, accessible, and non-invasive strategy to manage primary dysmenorrhea and its associated physical and psychological burdens in young women. The findings may have implications for broader implementation in university and workplace settings to support menstrual and general well-being.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 18 to 25 years
* Regular menstrual cycles (28 ± 7 days)
* History of primary dysmenorrhea for at least the past 6 months
* Menstrual pain intensity ≥40 mm on the Visual Analog Scale (VAS) during menstruation
* No history of childbirth
* Voluntarily agreed to participate and provided informed consent

Exclusion Criteria:

* History of pelvic surgery or pelvic pathology
* Use of hormonal treatments, contraceptives, or antidepressant medications
* Irregular menstrual cycles
* Pregnancy or history of childbirth
* Diagnosis of chronic pain due to other causes (e.g., fibromyalgia, endometriosis)
* Regular engagement in physical exercise or yoga practice in the past 3 months
* Any condition that may contraindicate moderate-intensity physical activity

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Primary dysmenorrhea is a condition that occurs in individuals with a uterus and regular menstrual cycles-thus, only biologically female participants were eligible.
Enrollment: 32 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Since the menstrual cycle length varies between 28-35 days Baseline, at the end of Menstrual Cycle 2 (approximately Day 56-70), and at the end of Menstrual Cycle 3 (approximately Day 84-105)
  Change in sleep quality assessed using the Sleep Diary across three menstrual cycles. Includes measures such as sleep onset latency, total sleep time, number of awakenings, and subjective sleep quality.
  Measure Type: Continuous (sleep parameters in minutes and Likert-scale scores) Sleep Onset Latency (in minutes) Total Sleep Time (in minutes) Number of Awakenings (count) Subjective Sleep Quality (Scale 1-5)
Aerobic Endurance | Since the menstrual cycle length varies between 28-35 days Baseline and at the end of Menstrual Cycle 3 (approximately Day 84-105)
  Change in aerobic endurance assessed via Incremental Shuttle Walk Test (ISWT) Measure Type: Continuous (distance in meters)
Aerobic Endurance | Since the menstrual cycle length varies between 28-35 days Baseline and at the end of Menstrual Cycle 3 (approximately Day 84-105)]
  Change in aerobic endurance assessed by Endurance Shuttle Walk Test (ESWT). Time to exhaustion during the ESWT, used to assess submaximal aerobic endurance Measure Type: Continuous (minutes)

SECONDARY OUTCOMES:
Menstrual Pain Intensity | Since the menstrual cycle length varies between 28-35 days Baseline, at the end of Menstrual Cycle 2 (approximately Day 56-70), and at the end of Menstrual Cycle 3 (approximately Day 84-105)
  . Pain severity will be assessed using a 100 mm Visual Analog Scale (VAS), where 0 mm indicates "no pain" and 100 mm indicates "worst imaginable pain." Measure Type: Continuous (VAS score in millimeters)Scores will be recorded during the first 3 days of menstruation across three menstrual cycles.
Menstrual Symptom Severity | Since the menstrual cycle length varies between 28-35 days Baseline and at the end of Menstrual Cycle 3 (approximately Day 84-105)
  Menstrual symptoms will be assessed using the Menstrual Symptom Questionnaire (MSQ), a 24-item self-report scale evaluating the severity and frequency of physical and emotional symptoms related to menstruation. The total MSQ score is calculated by summing item responses. Higher scores indicate worse (more severe) menstrual symptoms Measure Type: Continuous (total MSQ score) / Score range: 0 to 96

CONTACTS AND LOCATIONS:
Overall Officials: Seda Bicici Ulusahin, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and limitations in the consent obtained from participants.

REFERENCES:
- [Background] Super M. Can manifesting heterozygotes have cystic fibrosis? Thorax. 1999 Mar;54(3):194-5. doi: 10.1136/thx.54.3.194. No abstract available. PMID 10325892
- [Background] Freedman G. Buyers' guide to dental lasers. Lasers entering into the mainstream of dentistry. Dent Today. 2008 Dec;27(12):92, 94, 96 passim. No abstract available. PMID 19149046
- [Background] Bera TK, Rajapurkar MV. Body composition, cardiovascular endurance and anaerobic power of yogic practitioner. Indian J Physiol Pharmacol. 1993 Jul;37(3):225-8. PMID 8276501
- [Background] Divya TS, Vijayalakshmi MT, Mini K, Asish K, Pushpalatha M, Suresh V. Cardiopulmonary and Metabolic Effects of Yoga in Healthy Volunteers. Int J Yoga. 2017 Sep-Dec;10(3):115-120. doi: 10.4103/0973-6131.186162. PMID 29422741
- [Background] Lopes TR, Pereira HM, Bittencourt LRA, Silva BM. How much does sleep deprivation impair endurance performance? A systematic review and meta-analysis. Eur J Sport Sci. 2023 Jul;23(7):1279-1292. doi: 10.1080/17461391.2022.2155583. Epub 2022 Dec 15. PMID 36472094
- [Background] Aboagye E, Karlsson ML, Hagberg J, Jensen I. Cost-effectiveness of early interventions for non-specific low back pain: a randomized controlled study investigating medical yoga, exercise therapy and self-care advice. J Rehabil Med. 2015 Feb;47(2):167-73. doi: 10.2340/16501977-1910. PMID 25403347
- [Background] Rani M, Singh U, Agrawal GG, Natu SM, Kala S, Ghildiyal A, Srivastava N. Impact of Yoga Nidra on menstrual abnormalities in females of reproductive age. J Altern Complement Med. 2013 Dec;19(12):925-9. doi: 10.1089/acm.2010.0676. Epub 2013 May 6. PMID 23647406
- [Background] Sakuma Y, Sasaki-Otomaru A, Ishida S, Kanoya Y, Arakawa C, Mochizuki Y, Seiishi Y, Sato C. Effect of a home-based simple yoga program in child-care workers: a randomized controlled trial. J Altern Complement Med. 2012 Aug;18(8):769-76. doi: 10.1089/acm.2011.0080. Epub 2012 Jul 18. PMID 22808932
- [Background] Yang NY, Kim SD. Effects of a Yoga Program on Menstrual Cramps and Menstrual Distress in Undergraduate Students with Primary Dysmenorrhea: A Single-Blind, Randomized Controlled Trial. J Altern Complement Med. 2016 Sep;22(9):732-8. doi: 10.1089/acm.2016.0058. Epub 2016 Jun 17. PMID 27315239
- [Background] Chien LW, Chang HC, Liu CF. Effect of yoga on serum homocysteine and nitric oxide levels in adolescent women with and without dysmenorrhea. J Altern Complement Med. 2013 Jan;19(1):20-3. doi: 10.1089/acm.2011.0113. Epub 2012 Sep 10. PMID 22963270
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Iacovides S, Avidon I, Baker FC. What we know about primary dysmenorrhea today: a critical review. Hum Reprod Update. 2015 Nov-Dec;21(6):762-78. doi: 10.1093/humupd/dmv039. Epub 2015 Sep 7. PMID 26346058
- [Background] Dawood MY. Primary dysmenorrhea: advances in pathogenesis and management. Obstet Gynecol. 2006 Aug;108(2):428-41. doi: 10.1097/01.AOG.0000230214.26638.0c. PMID 16880317
- [Background] Ju H, Jones M, Mishra G. The prevalence and risk factors of dysmenorrhea. Epidemiol Rev. 2014;36:104-13. doi: 10.1093/epirev/mxt009. Epub 2013 Nov 26. PMID 24284871